CLINICAL TRIAL: NCT04104113
Title: HEalth-Related Quality of Life-intervention in Survivors of Breast and Other Cancers Experiencing Cancer-related Fatigue Using TraditionAL Chinese Medicine: The HERBAL Trial
Acronym: HERBAL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Collaborators: National Cancer Centre, Singapore (Other); Singapore Thong Chai Medical Institute (Unknown)
Responsible Party: Principal Investigator, Alexandre Chan, Associate Professor Dr. Alexandre Chan, National Cancer Centre, Singapore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIRB Ref. No: 2019/2135; TCMRG-3-NUS-01 (Other Grant/Funding Number: Ministry of Health Traditional Chinese Medicine Grant)
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Cancer; Fatigue; Cognitive Impairment
Keywords: Cancer; Cancer Related Fatigue; Cognitive Impairment; Survivorship; Traditional Chinese Medicine
MeSH Terms: conditions — Neoplasms; Fatigue; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XBYRT decoction (Experimental): Participants assigned to receive the modifed Xiang Bei Yang Rong Tang granules
  Interventions: Other: Modified Xiang Bei Yang Rong Tang
- Placebo (Placebo Comparator): Participants assigned to receive placebo (contains 5% of XBYRT) granules
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Modified Xiang Bei Yang Rong Tang — Modified Xiang Bei Yang Rong Tang is a combination of 15 herbal components and it is available in granules form to be dissolved in hot water for consumption
  Arms: XBYRT decoction
Other: Placebo — Placebo granules contain 5% XBYRT, colourant, bitterant and 95% starch filler
  Arms: Placebo

SUMMARY:
This study is a phase 2, randomized, double-blinded, placebo-controlled trial to evaluate the efficacy and safety of a Traditional Chinese Medicine decoction, the modified Xiang Bei Yang Rong Tang, in alleviating cancer related fatigue in cancer survivors.

DETAILED DESCRIPTION:
Cancer-related fatigue (CRF) is a distressing, persistent and subjective sense of physical, emotional, or cognitive tiredness related to cancer or its treatment. Currently there is a lack of effective conventional pharmacological intervention for treating this condition. Traditional Chinese Medicine (TCM) could be alternative therapy for managing CRF.

This study is a phase 2, randomized, double-blinded, placebo-controlled trial to examine the efficacy and safety of a TCM decoction, the modified Xiang Bei Yang Rong Tang (XBYRT) in alleviating CRF in cancer survivors. Study participants recruited from National Cancer Centre Singapore (NCCS) will be randomized to receive either the XBYRT or placebo decoction. Participants will take their assigned decoction daily for a duration of 8 weeks and will be assessed using patient reported outcome (PRO) questionnaires. PROs used are the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ 30) for QOL, the Multidimensional Fatigue Symptom Inventory Short Form (MFSI-SF) for fatigue and Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) Version 3 for cognitive abilities. The changes in scores measured by these assessment tools will be compared between the XBYRT intervention and placebo groups. Blood biomarkers such as inflammatory cytokines, mitochondrial DNA and oxidative stress markers will also be evaluated in the study participants. Additionally, adverse events or serious adverse events in participants will be monitored for safety.

Results from this study will provide a better understanding on the role of TCM in managing CRF.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥21 years
2. Clinically diagnosed cancer (Stages I-III)
3. Completed surgery/chemotherapy/radiotherapy for at least 1 month
4. At least one month after starting on aromatase inhibitors or ovarian suppression for breast cancer survivors
5. Not expected to receive surgery/chemotherapy/radiotherapy next 10 weeks
6. Fatigue screening score ≥4 for past 7 days
7. Life expectancy ≥3 months
8. Patients satisfy TCM syndrome differentiation as qi and blood deficiency Experience 2 major symptoms coupled with typical tongue and pulse conditions; 2 major symptoms and 1 possible symptom coupled with tongue and pulse conditions; 1 major symptom and at least 2 possible symptoms coupled with tongue and pulse conditions
9. Able to read and understand English or Mandarin

Exclusion Criteria:

1. Cancer recurrence and/or metastasis
2. Untreated co-morbidities causing fatigue (e.g. Severe anaemia, thyroid disorder)
3. On medications that cause fatigue (e.g. beta blockers)
4. Patients on warfarin
5. Cancer survivors receiving adjuvant therapy during the study period. Aromatase inhibitors and anti-HER2 monoclonal antibodies are acceptable.
6. Receiving or planning to receive treatment from other TCM practitioners during the study period
7. Breast feeding or intending to conceive/get pregnant during the study treatment period
8. Patients who present with yin deficiency and deficiency syndromes (e.g. phlegm-dampness, blood stasis, toxic-heat and qi stagnation)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2022-06-09 (Estimated)

PRIMARY OUTCOMES:
Difference in Global Health Status (GHS) score | 8 weeks from baseline
  Difference in Global Health Status (GHS) score from the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) between XBYRT interventional and placebo arms from baseline to 8 weeks after baseline. The GHS scale ranges in score from 0-100. A higher score represents a better quality of life

SECONDARY OUTCOMES:
Difference in Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF) scores | 4, 8 and 10 weeks from baseline
  Difference in MFSI-SF scores between XBYRT interventional and placebo arms. THE MFSI-SF consists of 30 items and has 5 subscales, each with 6 items: general fatigue, physical fatigue, emotional fatigue, mental fatigue, and vigour. The MFSI-SF measures different dimensions of fatigue, which can be combined to obtain an overall score. A higher score represents worse fatigue (total score ranges from -24 to 96)
Difference in Functional Assessment of Cancer Therapy-Cognitive (FACT-Cog) version 3 scores | 4, 8 and 10 weeks from baseline
  Difference in FACT-Cog V3 scores between XBYRT interventional and placebo arms. FACT-Cog v.3 will be used to assess subjective cognitive disturbances. These disturbances are assessed via 33 items in the domains of concentration, functional interference, mental acuity, memory, multitasking and verbal fluency (total score ranges from 0-148). A lower score represents worse cognitive function.
Incidence of adverse events | baseline, and 4, 8 and 10 weeks from baseline
  Adverse events reported according to the Adverse events Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Difference in EORTC QLQ-C30 version 3.0 Functional and Symptom scale scores | 4, 8 and 10 weeks from baseline
  Difference in EORTC QLQ-C30 scores between XBYRT interventional and placebo arms. The EORTC QLQ-C30 consists of 30 items across functional domains, symptoms domains and a global health status domain. All of the scales and single-item measures range in score from 0 to 100. A high score for a functional scale represents a high level of functioning. A high score for a symptom scale represents a high level of problems.
Mitochondrial DNA (mtDNA) content | baseline, 4, 8 and 10 weeks from baseline
  Mitochondrial DNA (mtDNA) content reduction in XBYRT interventional and placebo arms
Inflammatory cytokines : C reactive protein (CRP) and cytokines TNF-α, IL-1β, IL-6, and IL-8 | baseline, 4, 8 and 10 weeks from baseline
  Plasma inflammatory cytokine levels in XBYRT interventional and placebo arms
Oxidative stress markers : malondialdehyde (MDA), superoxide dismutase (SOD) and glutathione peroxidase (GSH-Px) | baseline, 4, 8 and 10 weeks from baseline
  Plasma oxidative stress markers levels in XBYRT interventional and placebo arms

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Chan, Pharm D, Principal Investigator — National University of Singapore, National Cancer Centre Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan A, Chan D, Ng DQ, Zheng HF, Tan QM, Tan CJ, Toh JHM, Yap NY, Toh YL, Ke Y, Wang ECA, Lim QPN, Ho HK, Chew L, Tan TJ. HEalth-Related Quality of Life-Intervention in Survivors of Breast and Other Cancers Experiencing Cancer-Related Fatigue and Associated Cognitive Symptoms Using TraditionAL Chinese Medicine: The 'HERBAL' Trial. Integr Cancer Ther. 2025 Jan-Dec;24:15347354251314514. doi: 10.1177/15347354251314514. PMID 39840742
- [Derived] Yap NY, Loo WS, Zheng HF, Tan QM, Tan TK, Quek LYP, Tan CJ, Toh YL, Ng CC, Ang SK, Tan VKM, Ho HK, Chew L, Loh KW, Tan TJY, Chan A. A study protocol for HEalth-Related quality of life-intervention in survivors of Breast and other cancers experiencing cancer-related fatigue using TraditionAL Chinese Medicine: the HERBAL trial. Trials. 2020 Nov 4;21(1):909. doi: 10.1186/s13063-020-04810-4. PMID 33187543